CLINICAL TRIAL: NCT04902573
Title: A Multicentre, Prospective, Non-interventional Trial Monitoring Therapy Pathways of Asthma Patients Treated With an Extrafine ICS/LABA/LAMA Single-inhaler Triple Therapy in a Real-world Setting and Characterizing the Effects on Health-related Out-comes
Brief Title: A Trial Monitoring Therapy Pathways of Asthma Patients Treated With an Extrafine ICS/LABA/LAMA Single-inhaler Triple Therapy in a Real-world Setting and Characterizing the Effects on Health-related Out-comes
Acronym: TriMaximize
Status: Completed | Type: Observational
Sponsor: Chiesi UK (Industry)
Collaborators: Gesellschaft für Therapieforschung mbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 548_TriMaximize; NIS 005 Pn (Other: International unique identifier (Chiesi)); 294788 (Other: IRAS)
Record Dates: First submitted 2021-05-17; First posted 2021-05-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Asthma
Keywords: Trimbow; asthma; triple therapy; beclometasone; formoterol; glycopyrronium; Trimaximize
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma patients: Trimbow pMDI prescribed for maintenance treatment of adult asthma as per the licensed indication.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — As this is a non-interventional trial, only data obtained within the current routine management of asthma at outpatient respiratory centres or GP centres will be documented.

SUMMARY:
TriMaximize, a non-interventional trial aims to collect prospective, longitudinal data from asthma patients under routine care, for whom their treating physician has decided to prescribe Trimbow® (beclometasone/formoterol/glycopyrronium).

DETAILED DESCRIPTION:
TriMaximize, a non-interventional trial aims to collect prospective, longitudinal data from asthma patients under routine care, for whom their treating physician has decided to prescribe Trimbow® (beclometasone/formoterol/glycopyrronium).

Trimbow is a fixed triple therapy containing a long-acting muscarinic antagonist (LAMA, glycopyrronium), a long-acting beta-adrenergic agonist (LABA, formoterol) and an inhaled corticosteroid (ICS, beclometasone).

Asthma patients often need to use multiple inhalers as part of their therapy, which require different inhalation techniques. It has been shown that the use of several inhalers of different mode of action, design and dosage requirements may have a detrimental effect on patient adherence and subsequent treatment outcomes.

In this prospective, non-interventional trial, the investigators aim to evaluate aspects of adherence to Trimbow, a single-inhaler triple therapy (SITT) as a maintenance treatment of asthma, to gather knowledge from routine care on whether appropriate step-up to SITT leads to greater adherence and better health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age,
2. Patients with confirmed leading diagnosis of asthma with or without concomitant COPD,
3. Physician decision to start fixed triple therapy with ICS/LABA/LAMA (Trimbow MS or HS) according to its current authorised indication. The treatment decision must be made independently from participation in this NIS,
4. Patients willing and able to sign an informed consent for use of their pseudonymised clinical data within the present non-interventional study.

Exclusion Criteria:

1) Participation in an interventional clinical trial within 30 days prior to enrolment into the present non-interventional study or planned enrolment in an interventional clinical trial during the observational period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will only be included in the Non-Interventional Trial if Trimbow® has been prescribed in line with its current marketing authorisation and the guidance specified in the summary of product characteristics (SmPC).
  Physicians are urged to offer enrolment to all of their eligible patients consecutively as they present for their routine visit, and not select patients from their patient database.
  Eligible patients may only be included in the NIT after providing written (witnessed, where required by law or regulation), IEC-approved informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
To describe patient characteristics and therapy pathways for patients with a diagnosis of moderate to severe asthma who are treated with Trimbow in real world practice | 12 months
  Descriptive analysis of patient demographics

SECONDARY OUTCOMES:
Assess asthma control (ACT) | 12 months
  Change from baseline in ACT scores
Assess quality of life | 12 months
  Change from baseline in Mini-AQLQ scores
Assess treatment adherence | 12 months
  Change from baseline in TAI scores
Analyse parameters of lung function using spirometry | 12 months
  Change from baseline in FEV1
Analyse parameters of small airways disease | 12 months
  Change from baseline in small airway function measured by pre-dose AUCAX (Area under the curve of reactance) using available oscillometry system
Analyse parameters of asthma-related airway inflammation | 12 months
  Change from baseline in percentage of patients with a fraction of exhaled nitric oxide (FeNO) below or above 20 ppb
Analyse parameters of persistent airflow limitation | 12 months
  Change from baseline in percentage of patients with persistent airflow limitation (PAL); PAL defined as post-BD FEV1 <80% predicted and post-BD FEV1/FVC Ratio < 0.7
Analyse the incidence of asthma exacerbations | 12 months
  Number of exacerbations 12 months prior to baseline and during study
Analyse the severity of asthma exacerbations as defined by the American Thoracic Society/European Respiratory Society (ATS/ERS) classification of asthma exacerbations | 12 months
  Severity of exacerbations, defined according to the ATS/ERS classification of asthma exacerbations, will be analysed 12 months prior to baseline and during study
Analyse use of rescue medication | 12 months
  Use of any rescue medication 7 days prior to baseline and during study 7 days prior to respective visit
Analyse use of systemic corticosteroids | 12 months
  Use of any systemic corticosteroids 12 months prior to baseline and during study
Assess adverse events associated with use of Trimbow | 12 months
  Assessment of the number and type of adverse events
Assess retention rate with Trimbow | 12 months
  Assess continuation of treatment with Trimbow (retention rate of Trimbow) at month 12

CONTACTS AND LOCATIONS:
Overall Officials: Richard Russell, PhD, MBBS, Principal Investigator — University of Oxford
Locations (1):
- The Haven Surgery, The Haven, Burnhope,, Durham, County Durham, United Kingdom

IPD SHARING:
Plan to Share IPD: No